CLINICAL TRIAL: NCT00619580
Title: Ampicillin-sulbactam Resistant E.Coli at UPMC
Status: Withdrawn | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO08010298
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Positive E Coli Infections
Keywords: E coli
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- positive E coli: positive E coli at UPMC

SUMMARY:
The information collected will optimize the management of patients with gram negative bacteremia. Approximately 300 patients with Gram negative bacteremia are cared for each year at UPMC-P. Published medical literature suggests that mortality from this infection exceeds 20%. The aim of this research is to determine the risk factors for bacteriologic failure of antibiotic therapy, risk factors for antibiotic resistance in bloodstream isolates and risk factors for mortality from Gram negative bacteremia. Modifiable risk factors can then be tackled by a future interventional study.

DETAILED DESCRIPTION:
The information collected will optimize the management of patients with gram negative bacteremia. Approximately 300 patients with Gram negative bacteremia are cared for each year at UPMC-P. All sites are collecting the following information that was collected as part of the patient's clinical treatment. The following variables will be collected at all sites: time and location of positive cultures, underlying diseases and severity of illness, recent immunomodulative therapies, physical exam findings, laboratory and radiographical data, antimicrobial usage within 14 days of onset of bacteremia, microbiological data and resistance patterns, choice of antibiotics once organism identified, suspected source of bacteremia, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome,gender, height, weight, ethnicity, and past medical history (please see attached clinical data collection worksheet dated 4/2005). We will also collect information retrospectively for one year and prospectively for one year. The bacteria in the patient's blood cultures will be subcultured (after the diagnosis has been obtained since the microbiology lab would otherwise destroy the culture) and provided to the honest broker who will deidentify the specimen and link it to the medical information collected (which will also be deidentified by the honest broker). The following evaluation will be performed on these samples. The minimal inhibitory concentration of the antibiotic used in treatment will be performed by the E-Test method (AB Biodisk, Solna, Sweden). Specific mechanisms of antimicrobial resistance will be studied with emphasis on the presence of beta-lactamases produced by the bacteria. This evaluation will be performed by analytical isoelectric focusing techniques as well as PCR and gene sequencing analysis to determine genes encoding beta-lactamases. Biologic samples will be under the control of the principal investigator of this research project. All samples provided to the investigators are deidentified by the honest broker and will be coded with numbers. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location that only the honest broker has access to. The investigators on this study will keep the samples indefinitely. Samples will be kept in the investigator's laboratory located in Scaife Hall, room 812, 3500 Terrace Street. At no time with the research investigators have access to any patient identifers. Medical record information and bacteria samples from facilities outside of UPMC will be provided to the PI de-identified. At not time will the anyone on the research team have access to patient identifiers. All information and bacteria are collected as part of the patient's clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients at the aforementioned institutions that have Gram negative bacteremia will be included in the study.
* Women with childbearing potential will also be included in this study. Since this is an observational study, no added risk is conferred to the woman or potential progeny. HIV serostatus will not be specifically investigated for participation in this study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: E coli positive infections at UPMC
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The aims of this study are to: Determine the risk factors for multidrug resistance (ESBL production) in bloodstream isolates of Gram negative bacilli, | 5 years

SECONDARY OUTCOMES:
determine the risk factors for failure of prompt clearance of the blood of Gram negative bacteria | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yohei Doi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States